CLINICAL TRIAL: NCT03032341
Title: Mobility Assessment Using Surrogates in Elderly Participants
Acronym: MAT
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Sunghye Kim, Assistant Professor, Wake Forest University Health Sciences
Other Study IDs: IRB00040417
Record Dates: First submitted 2017-01-18; First posted 2017-01-26 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Mobility Limitation
Keywords: mobility assessment tool
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: 20 patient in poor mobility group (MAT-sf < 51.38 in men and <45.61 in women), mid-mobility group (51.38< MAT-sf≤65.5 in men and 45.61≤MAT-sf<54.02) and high mobility group (MAT-sf>65.5 in men and MAT-sf>54.02 in women) for a total of 60 patients.
- Surrogate group: A family member/caregiver that attends visits with the patient and will be asked to answer the Mobility Assessment Test questionnaire on behalf of the patient at the initial visit and the follow up visit 1-14 days later.

SUMMARY:
The purpose of this research study is to find out if mobility (the ability to move around) can be reliably assessed by having the family or care giver caregiver take a video based test for the patient. If this study shows that mobility can be assessed by family or caregiver, this information can be used in situations where mobility cannot be measured directly in patients. A total of 60 patients and 60 family/caregivers at Wake Forest Baptist Medical Center will take part in this study. Patients physical function will be assessed using a test that uses short movie clips to assess mobility. Patients will be asked to watch ten short (~10 seconds each) movie clips that describe various tasks such as climbing up hills or walking and estimate if they can perform the tasks. The familymember/caregiver will be also asked to answer the questions on behalf of the patient. The family member/caregiver will be asked to return to take the same test in the next 1-14 days. The patient will be in the study for one day. There is no intervention, this is observational.

DETAILED DESCRIPTION:
According to the U.S. Census Bureau projections, the number of persons 65 years of age or older will increase from roughly 40 million in the year 2010, to 88.5 million in 2050, a net increase of 121%. During this same time period, the number of persons 85 years of age or older will increase by 227%; accounting for nearly 5% of the U.S. population. Mobility and functional status are important predictors of outcomes in this rapidly growing elderly population. It has shown that walking speed and physical function, measured by Short Physical Performance Battery (SPPB) are predictors of mortality in community-dwelling older men and women. It was also reported that gait speed predicts incident disability in community dwelling elderly subjects. In our prior study, we have demonstrated that, mobility, assessed using an animated video clip based assessment tool, Mobility Assessment Tool-short form (MAT-sf) predicts postoperative complications, length of stay and nursing home placement in elderly patients (>69) who were undergoing elective surgery that requires overnight hospitalization and more clinical practices use physical function and mobility as a tool to predict outcomes.

However, these assessments are not always readily available, especially in clinical situations when acute illnesses or injuries occurred without any chance to assess the baseline status, such as acute myocardial infract, rapidly progressing sepsis or catastrophic trauma. In these cases, patients are often sedated, intubated, have altered mental status, or too unstable to perform even non-invasive testing. Although some clinicians or researchers feel that surrogate can accurately assess the patients' baseline physical function and mobility status, it was never been tested.

The investigators hypothesize that mobility assessment done on surrogates, using MAT-sf will have high compatibility with the assessment done on elderly patients. Surrogates are defined as a person who spends >2 hours a day or 8 hours a week with the patient and accompany the patient to most of their medical appointments. The investigators will test the hypothesis at the Preoperative Assessment Clinic since this clinic sees high volume of elderly patients and patients at this clinic tend to have their caregiver with them during the appointments.

Investigators will enroll 20 patients in poor mobility group (MAT-sf < 51.38 in men and <45.61 in women), 20 patients into the mid-mobility group (51.38< MAT-sf≤65.5 in men and 45.61≤MAT-sf<54.02) and 20 patients into the high mobility group (MAT-sf>65.5 in men and MAT-sf>54.02 in women) for a total of 60 patients and one surrogate per patient for a total of 120 unique participants.

To assess mobility, participants will be instructed on the use of the Mobility Assessment Tool-short form (MAT-sf). The MAT-sf is a 10-item computer based assessment of mobility using animated video clips. The 10 items in the MAT-sf cover a broad range of functioning. The items include walking on level ground, a slow jog, walking outdoors on uneven terrain, walking up a ramp with and without using a handrail, stepping over hurdles, ascending and descending stairs with and without the use of a handrail, and climbing stairs while carrying bags. The items were previously selected based on individual response and information curves derived from Item Response Theory. Each item is accompanied by an animated video clip together with the responses for that question (number of minutes, number of times, yes/no). The test will be performed on an I-PAD and scores will be saved to an exportable file. The time required to do the test with instructions from the examiner is expected to be no longer than 5 minutes. While the patient is completing the MAT-sf assessment, the surrogate will be directed to a separate room to complete MAT-sf for the patient ("Do you think Mr ** can climb up this hill?) , so there is no interaction between the patient and the surrogate during the assessment. Investigators will measure the compatibility between patients-surrogates mobility using MAT-sf and will also assess the stability of surrogate MAT-sf.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 years and older being seen at the PAC;
* Patients who have caregiver or family who meet the criteria for surrogate as above;
* Patients scheduled for elective surgical procedures.

Exclusion Criteria:

* Patients who have a language barrier which will prohibit them from understanding the questionnaire and directions connected to the use of the MAT-sf;
* Patients who are not able to sign their own surgical consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 60 patients being seen in the post operative assessment clinic will be asked to complete the Mobility Assessment Tool. A family member/caregiver of each patient will be asked to complete the test on the behalf of the patient at the same visit and asked to complete again 1-14 days later.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
Change in MAT-sf score between patients and surrogates | 1-14 days
  Investigators will measure the compatibility between patients-surrogates mobility using MAT-sf.

CONTACTS AND LOCATIONS:
Overall Officials: Sunghye Kim, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No